CLINICAL TRIAL: NCT03904719
Title: Combination of CM082 With JS001 in Patients With Advanced Small-cell Lung Cancer (SCLC) Who Progressed on First-line Treatment: a Phase II Study
Brief Title: CM082 and JS001 in Patients With Advanced Small-cell Lung Cancer (SCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-II-203
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — vorolanib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 plus JS001 (Experimental): CM082 tablets 150mg is orally given once daily in a 28-day cycle, combinational JS001 240mg was given intravenously on day 1 once every 21 days.
  Interventions: Drug: CM082 plus JS001

INTERVENTIONS:
Drug: CM082 plus JS001 — CM082: 150mg once a day orally (taken within half an hour after breakfast) JS001: An intravenous infusion of a solution having a concentration of 1-3mg/ml was prepared with 0.9% physiological saline, and administered once every three weeks. Using an inline filter (0.2 or 0.22 μm), the drug was diluted with physiological saline and intravenously administered within 60 minutes.
  Other Names: Vorolanib; Toripalimab

SUMMARY:
This study was a single-arm, multi-center, phase II study, which is aimed to evaluate the efficacy and safety of CM082 combined with JS001 as the second-line treatment of advanced small cell lung cancer. Eligible patients will receive CM082 tablets 150mg once daily orally in combination with JS001 (240mg, intravenously) every 21 days. Treatment continues until disease progresses , intolerable toxicity, or withdraw.

DETAILED DESCRIPTION:
This study was a single-arm, multi-center, phase II study, which is aimed to evaluate the efficacy and safety of CM082 combined with JS001 as the second-line treatment of advanced small cell lung cancer. Eligible patients will receive CM082 tablets 150mg once daily orally in combination with JS001 (240mg, intravenously) every 21 days. Treatment continues until disease progresses , intolerable toxicity, or withdraw.

The primary endpoint is tumor response per investigator assessment according to response evaluation criteria in solid tumors (recist) version 1.1, secondary endpoints include disease control rate, progression-free survival, overall survival, safety and tolerability. iRECIST is also implemented for tumor response assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent, inoperable, metastatic SCLC (stage III/IV period);
* Progressive disease after prior standard systemic treatment;
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1;
* Life expectancy of at least 12 weeks;
* At least one measurable lesion according to the RECIST 1.1;
* Adequate organ functions;
* Negative serum pregnancy test results within 7 days prior to the first dose of the study drug;
* Patients willing to obey the schedule for study and follow-up procedures;
* Patients who can understand the nature of the study and sign voluntarily the informed consent.

Exclusion Criteria:

* Patients who have previously received treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or VEGFR TKI therapy (sunitinib, sorafenib, pizopren, axitinib, bevacizumab, remomituzumab, nidanib, vandetanib, etc), or CTLA-4 inhibitor (Ipilimumab, etc).
* Patients who are presently receiving other systematic antitumor therapies.
* Patients who developed other malignancies (not including cured basal cell tumor of skin, endoscopically resected early gastrointestinal tract [GI] tumor, and cervical carcinoma in situ) except lung cancer in the past 2 years.
* Patients receiving a major surgery or immunotherapy in the past 4 weeks prior to the first dose; and patients receiving a radiotherapy within 2 weeks prior to the first dose.
* Patients with brain metastases or meningeal metastases.
* Have received hematopoietic stimulating factors within 1 week prior to the first dose of the study drug.
* Patients who previously received stem cell transplantation or organ transplantation.
* Patients with swallowing dysfunction, active gastrointestinal disease, or other disorders that may influence significantly absorption, distribution, metabolism, or excretion of CM082.
* Patients with active hepatitis B, hepatitis C virus antibody positive , HIV antibodies, or treponema pallidum antibody positive.
* Patients with a prior history of interstitial lung disease, history of drug-induced interstitial lung disease, history of radiation pneumonia requiring a steroid therapy, or any clinical indications for active interstitial lung disease.
* Patients who are known to be allergic to JS001 or CM082 or any excipients of the study drugs.
* Patients receiving in the past 14 days or requiring concurrently the following drugs during treatment: Drugs that may result in a risk for QTc prolongation and/or torsades de pointes; or CYP3A potent inhibitors or potent inducers.
* Patients with other severe, acute or chronic medical conditions (including incontrollable diabetes mellitus, or medical disease or mental disease, or laboratory test abnormality) that may increase study-related risk or may interfere with interpretation of the research results, in the viewpoints of the investigator.
* Patients with other conditions that not suitable to participate in this study, as considered by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  The proportion of patients with complete remission (CR) and partial remission (PR) in all patients. Disease progression will be evaluated according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  The internal between the date of enrollment and the date of disease progression, unaccepted toxicity, or death according to RECIST 1.1 and iRECIST.
Overall survival | 36 months
  The internal between the date of randomization and the date of death
Disease Control Rate | 6 months
  The proportion of patients with complete remission (CR), partial remission (PR) and stable disease (SD) in all patients. Disease progression will be evaluated according to RECIST 1.1 and iRECIST.
Duration of Response | 12 months
  The time between patients's first time to complete or partial remission to disease progression.
Time to response | 12 months
  The internal between the date of enrollment and the date of documented tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Study Chair — National Cancer Center/Cancer Hospital
Locations (2):
- China (2):
  - National Cancer Center/Cancer Hospital, Beijing
  - The First Hospital of China Medical University, Shenyang